CLINICAL TRIAL: NCT04791657
Title: Factors Associated With Postoperative Complications After the Surgical Treatment of Appendicitis in Elderly Patients
Brief Title: Outcome of Elderly Patients With Appendicitis
Status: Completed | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suleyman Utku Celik, Principal Investigator, Gulhane Training and Research Hospital
Other Study IDs: Gulhane2021-51
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Appendicitis Acute
Keywords: appendicitis; geriatrics
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without complications: Patients with uneventful recovery
  Interventions: Procedure: Appendectomy
- Patients with complications: Patients experiencing complications within 30 days postoperatively
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Surgical treatment for appendicitis

SUMMARY:
This study aims to evaluate factors that predict 30-day complications after the surgical treatment of appendicitis in elderly patients.

DETAILED DESCRIPTION:
Appendicitis in elderly patients is more challenging due to delayed presentation and higher comorbidities, which is associated with increased postoperative morbidity and mortality. In this study, we aim to investigate the factors that predict 30-day complications after the surgical treatment of appendicitis in elderly patients. Records of patients who underwent appendectomy for appendicitis will be extracted. The primary outcome is 30-day postoperative complications. Independent variables examined include demographics, comorbidities, preoperative laboratory values, pathological findings, and surgical features. Both univariate and multivariate regression will be performed to identify factors associated with postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Patients undergoing appendectomy for acute appendicitis (pathologically confirmed)
* Patients having complete records of clinical data and postoperative follow-up records

Exclusion Criteria:

* Patients younger than 65 years
* Patients undergoing an appendectomy as part of another major operation or those with appendiceal malignancy
* Patients who are treated nonoperatively for acute appendicitis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 65 years and older undergoing appendectomy for acute appendicitis are included in this study
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
30-day postoperative complication rate | 30 days
  The primary clinical outcome of interest is 30-day postoperative complications. The Clavien-Dindo classification will be used to grade postoperative outcomes and complications

SECONDARY OUTCOMES:
In-hospital mortality rate | 30 days
  In-hospital mortality is defined as death occurring during the hospital stay after the surgical procedure
30-day readmission rate | 30 days
  30-day readmission is defined as unplanned readmission to the hospital within 30 days of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman U Celik, MD, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Angeramo CA, Dreifuss NH, Giacone J, Schlottmann F. Outcomes of Acute Appendicitis in Elderly Patients: a Single Center Analysis of 2000 Laparoscopic Appendectomies. J Gastrointest Surg. 2020 Dec;24(12):2859-2861. doi: 10.1007/s11605-020-04726-z. Epub 2020 Aug 31. No abstract available. PMID 32865733
- [Background] Yang J, Yu K, Li W, Si X, Zhang J, Wu W, Cao Y. Laparoscopic Appendectomy for Complicated Acute Appendicitis in the Elderly: A Single-center Experience. Surg Laparosc Endosc Percutan Tech. 2017 Oct;27(5):366-368. doi: 10.1097/SLE.0000000000000447. PMID 28708770
- [Background] Hui TT, Major KM, Avital I, Hiatt JR, Margulies DR. Outcome of elderly patients with appendicitis: effect of computed tomography and laparoscopy. Arch Surg. 2002 Sep;137(9):995-8; discussion 999-1000. doi: 10.1001/archsurg.137.9.995. PMID 12215147
- [Background] Pokharel N, Sapkota P, Kc B, Rimal S, Thapa S, Shakya R. Acute appendicitis in elderly patients: a challenge for surgeons. Nepal Med Coll J. 2011 Dec;13(4):285-8. PMID 23016482